CLINICAL TRIAL: NCT04790929
Title: Assessing the Effects of the Muse Meditation System on Cognition and Well-being
Acronym: MuseCog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: InteraXon, Inc. (Industry); Cambridge Brain Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 118280
Record Dates: First submitted 2021-03-01; First posted 2021-03-10 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Change

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular Muse Meditation System - No Coaching (Experimental): Participants will join a 1.5-hour virtual onboarding session where they will complete their first Muse session. Participants will then be asked to use the Muse Meditation system for a minimum of 5 minutes a day (in one or multiple sessions), a minimum of 5 days a week, for 6 weeks. If they wish to use the system more frequently within the 6 weeks, they will be encouraged to do so and will be able to choose between all the styles of meditation available in the Muse Meditation System (Mind, Heart, Breath, Body, Guided or Sleep Journeys). For any challenges that arise, participants will have unlimited access to Muse Customer Care via phone, email, and video where appropriate during normal business hours.
  Interventions: Device: Muse
- Regular Muse Meditation System - Additional Coaching (Experimental): The procedure will be identical to Group 1 above, but in addition, all participants will be asked to join regular online coaching sessions. Participants will be divided into 8 cohorts of 10 people per cohort. Each cohort will be offered group coaching once per week. Coaches will be versed in Mindfulness and how to use Muse. Coaching will take place virtually using Interaxon's Zoom account. Throughout the coaching, all participants will be referred to via their first names or their anonymized login names. In addition, for any challenges that arise, participants will have unlimited access to Muse Customer Care via phone, email, and video where appropriate during normal business hours.
  Interventions: Device: Muse; Behavioral: Meditation Coaching
- Controls (No Intervention): The participants in the control group will receive a Muse Device, which they will be free to keep at the end of the study. They will be asked not to open and/or use the Muse device until the entire study is complete. On day 1 of the Study, they will complete the Cambridge Brain Sciences online cognitive assessment battery, plus a longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness, anxiety and depression and sleep quality. At the completion of the study controls will be offered optional, free group coaching sessions if they complete the study requirements.

INTERVENTIONS:
Device: Muse — Interaxon markets a head-worn EEG biofeedback device ('Muse') to encourage and aid effective meditation and sleep. This device has been previously shown to improve workplace wellness, fatigue and quality of life, and performance on the Stroop Task. It has also been shown to improve physiological markers associated with improved relaxation. Muse has been shown to have an EEG signal comparable to a clinical grade EEG.
  Arms: Regular Muse Meditation System - Additional Coaching; Regular Muse Meditation System - No Coaching
Behavioral: Meditation Coaching — Participants will be asked to use the Muse Meditation system for a minimum of 5 minutes a day (in one or multiple sessions), a minimum of 5 days a week, for 6 weeks and will be coached in how to do so. Coaches will be versed in Mindfulness and how to use Muse. Coaching will take place virtually using Interaxon's Zoom account.
  Arms: Regular Muse Meditation System - Additional Coaching

SUMMARY:
Interaxon markets a head-worn EEG biofeedback device ('Muse') to encourage and aid effective meditation and sleep. This device has been previously shown to improve workplace wellness, fatigue and quality of life, and performance on the Stroop Task. It has also been shown to improve physiological markers associated with improved relaxation. What is not known, is whether the use of the Muse devices can improve cognitive function. In this study, the investigators will examine whether use of the Muse Meditation system by healthy participants, leads to improvements in cognition, sleep quality, mindfulness, improvement in quality of life scores, reduction in perceived stress levels, and improvement in cognitive markers relevant for safety and increased success in the workplace.

DETAILED DESCRIPTION:
Meditation is a non-invasive technique that has recently gained significant popularity for its ability to effect positive change on the mind and body. Even a brief (4 sessions) meditation training intervention has been shown to lead to improvements in various areas of cognitive function [1], stress and anxiety, and it has been shown to improve sleep in older adults better than a sleep hygiene course [2]. Mindfulness is now being extensively used in the workplace to promote various aspects of workplace wellness [3], and workplace health and safety [4].

Interaxon markets a head-worn EEG biofeedback device ('Muse') to encourage and aid effective meditation and sleep. This device has been previously shown to improve workplace wellness, fatigue and quality of life, and performance on the Stroop Task. It has also been shown to improve physiological markers associated with improved relaxation.

In this study, the investigators will examine whether use of the Muse Meditation system by healthy participants, leads to improvements in cognition, sleep quality, mindfulness, improvement in quality of life scores, reduction in perceived stress levels, and improvement in cognitive markers relevant for safety and increased success in the workplace.

240 participants will be randomly divided into 3 groups with 80 participants in each group (see below).

Group 1 will use the Muse Meditation system with no coaching.

Group 2 will use the Muse Meditation system with additional online coaching.

Group 3 will be a control group and will not use any of the Muse Meditation systems

On day 1 of the Study, all participants will complete the Cambridge Brain Sciences online cognitive assessment battery, plus a longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness and sleep quality. They will then begin the 6-week study according to their following Group assignments:

Group 1: Regular Muse Meditation System - No Coaching:

Participants will join a 1.5-hour virtual onboarding session where they will complete their first Muse session. Participants will then be asked to use the Muse Meditation system for a minimum of 5 minutes a day (in one or multiple sessions), a minimum of 5 days a week, for 6 weeks. If they wish to use the system more frequently within the 6 weeks, they will be encouraged to do so and will be able to choose between all the styles of meditation available in the Muse Meditation System (Mind, Heart, Breath, Body, Guided or Sleep Journeys). For any challenges that arise, participants will have unlimited access to Muse Customer Care via phone, email, and video where appropriate during normal business hours.

Group 2: Regular Muse Meditation System - Additional Coaching The procedure will be identical to Group 1 above, but in addition, all participants will be asked to join regular online coaching sessions. Participants will be divided into 8 cohorts of 10 people per cohort. Each cohort will be offered group coaching once per week. Coaches will be versed in Mindfulness and how to use Muse. Coaching will take place virtually using Interaxon's Zoom account. Throughout the coaching, all participants will be referred to via their first names or their anonymized login names. In addition, for any challenges that arise, participants will have unlimited access to Muse Customer Care via phone, email, and video where appropriate during normal business hours.

Group 3: Controls The participants in the control group will receive a Muse Device, which they will be free to keep at the end of the study. They will be asked not to open and/or use the Muse device until the entire study is complete. On day 1 of the Study, they will complete the Cambridge Brain Sciences online cognitive assessment battery, plus a longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness, anxiety and depression and sleep quality. At the completion of the study controls will be offered optional, free group coaching sessions if they complete the study requirements.

At the end of Week 6 (at the completion of the main study period), all participants will be reassessed using the Cambridge Brain Sciences online cognitive assessment battery , and the longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness and sleep quality.

All participants will also complete a brief debriefing questionnaire at the end of Week 6, reporting their experiences about the study.

They will again be assessed using the Cambridge Brain Sciences online cognitive assessment battery, and the longer questionnaire about stress levels, workplace wellness, quality of life, mindfulness and sleep quality at the end of Week 12 (6 weeks after completing the main study period).

Hypothesis 1: Using the Muse Meditation system for 6 weeks will yield improvements in cognitive performance on the Cambridge Brain Sciences battery, improvements in self-reported sleep quality (e.g. decreased latency to sleep, improved sleep duration), improvements on measures of mindfulness, improvement in quality of life scores, reduction in perceived stress levels, reduction in anxiety, and improvement in cognitive markers (derived from the Cambridge Brain Sciences scores) relevant for safety and increased success in the workplace. The investigators expect to see these changes in both experimental groups relative to the control group.

Hypothesis 2: These changes will persist well beyond the period of the study and will be detectible at the 12-week follow-up session.

Hypothesis 3: The participants who use the Muse Meditation system and have additional coaching (Group 2), will experience improvements in cognition, stress, anxiety, and other quality of life measures over and above those experienced by those who use the Muse Meditation system with no coaching (Group 1).

ELIGIBILITY:
Inclusion Criteria:

The study will be open only to all Hatch Inc employees in Canada.

Exclusion Criteria:

If participants do not own a smart phone

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Cognition | 12 weeks
  The primary outcome will be scores on the Cambridge Brain Sciences (CBS) cognitive battery The Cambridge Brain Sciences (CBS) battery assesses aspects of memory, attention, planning, and reasoning, using a web-based interface that can be self-administered at home through any internet browser.

SECONDARY OUTCOMES:
Perceived Stress Scale | 12 weeks
  Quality of life will be scoresd on self-reported Perceived Stress Scale.
Anxiety Questionnaire | 12 weeks
  Anxiety will be scored using General Anxiety Disorder 7 Scale
Depression Questionnaire | 12 weeks
  Depression will be measured using will be scored using Patient Health Questionnaire 9

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Canada

IPD SHARING:
Plan to Share IPD: Undecided